CLINICAL TRIAL: NCT05748886
Title: Global Cohort Study: Hernias, Pathway and Planetary Outcomes for Inguinal Hernia Surgery
Brief Title: A Global Prospective Study on Inguinal Hernia Surgery
Acronym: HIPPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: HIPPO
Record Dates: First submitted 2023-02-08; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Inguinal Hernia; Groin Hernia; Surgery
Keywords: Inguinal; Hernia; Inguinal Hernia; Groin Hernia; Audit; Groin hernia management; mesh repair; non-mesh repair; laparoscopic repair; Global Surgery; Surgery
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Period 1: 00:00 30th Jan 2023 - 23:59 26th Feb 2023 (+ 30 Day Follow-up)
- Period 2: 00:00 27th Feb 2023 - 23:59 26th Mar 2023 (+ 30 Day Follow-up)
- Period 3: 00:00 27th Mar 2023 - 23:59 23th Apr 2023 (+ 30 Day Follow-up)
- Period 4: 00:00 24th April 2023 - 23:59 21st May 2023 (+ 30 Day Follow-up)

SUMMARY:
The primary aim of the HIPPO study is to identify compliance to audit standards (pre-operative and intraoperative) standards for the repair and management of inguinal hernia.

A prospective, multicentre, cohort study will be delivered by NIHR Unit on Global Surgery globally. Mini-teams of up to five collaborators per data collection period will prospectively collect data over a continuous 28-day period at each participating centre. This will be on consecutive patients undergoing elective and/or emergency primary inguinal hernia surgery, with follow-up to 30 postoperative days.

DETAILED DESCRIPTION:
Inguinal hernia surgery is one of the most common elective operations around the world. It was significantly down-prioritised during the pandemic, with fewer planned procedures and a likely increase in a global backlog. According to the most updated data, there are 74,822 patients waiting for inguinal hernia repair in the United Kingdom's National Health Service (NHS), although the recommended expected waiting time should not exceed 18 weeks. It is likely that other countries face the same problem, although such granular data does not exist. Additionally, while waiting for an elective repair, complications of inguinal hernia might arise and an emergency surgery might be needed. Identifying the scale of the global backlog at a global level will inform policy makers on the best strategies to optimise this elective surgical pathway.

Different surgical techniques exist, with different mesh and non-mesh techniques being described. The most up-to-date international guidelines recommend Lichenstein as the gold-standard for open repair of inguinal hernias, but a more tailored approach is recommended. The patient, the hernia type, and the surgeon's expertise will influence the choice of surgical technique which leads to a wide variation worldwide. Additionally, in areas where there is a deficit of surgeons, task sharing and task shifting might be implemented. Identification of this practice across the world and the outcomes associated with it will inform future research in this area.

Finally, as inguinal hernia repair is a very common procedure, it can reflect the global uptake of environmentally sustainable measures in elective surgery. Achieving a net zero health system is only possible if reducing the carbon output from operating theatres is included. Different countries might have different protocols and measures adopted to be environmentally sustainable that could be used in different settings. Understanding the baseline point of these practices is extremely important to inform future studies in this area.

ELIGIBILITY:
Inclusion Criteria:

Summary: Consecutive patients during the selected study period undergoing elective or emergency primary inguinal hernia repair through any operative approach.

Inclusion criteria:

* Age: Paediatric and adult patients
* Procedure: Primary inguinal hernia repair, where this is the main procedure. For patients with bilateral inguinal hernias, data should be entered only for the larger of the two.
* Approach: Open groin incision, laparoscopic, laparoscopic assisted, laparoscopic converted, robotic, robotic converted procedures are all eligible. Patients with open incisions other than groin incision (e.g. laparotomy) are excluded.
* Urgency: Patients undergoing planned (elective) surgery or emergency surgery

Exclusion Criteria:

Procedures:

* Recurrent inguinal hernias
* Surgeries where inguinal hernia repair is not the main procedure, but performed as an additional procedure (eg patient operated for colon cancer and undergoing inguinal hernia repair during the same operation).
* If patients are undergoing repair of two different types of hernia they can be included if the inguinal hernia repair is the main operation. (e.g. patient undergoing both inguinal and umbilical hernia repair). However, if the inguinal hernia repair is a secondary procedure to a larger non-inguinal hernia repair, patients should be excluded (e.g patient undergoing both large incisional hernia repair and inguinal hernia repair).
* Laparoscopic converted to open midline procedures
* Patients undergoing surgery with intent of repair of inguinal hernia, where no hernia inguinal hernia was identified (e.g. intra-operative findings of adenopathy, femoral hernia, obturator hernia)

Return to theatre:

* Each individual patient should only be included in the study once. Patients returning to theatre due to complications following earlier surgery can only be included if their index procedure has not already been included in the HIPPO audit.
* Patients with bilateral hernias undergoing repair with two separate procedures in two different times, should only be included for the first procedure.

Data should be collected on consecutive patients operated at each centre during the data collection period. This means that all eligible patients should be included.

Strategies to identify consecutive eligible patients could include:

* Daily review of elective theatre lists.
* Daily review of handover sheets and ward lists.
* Daily review of theatre logbooks (both elective).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients during the selected study period undergoing elective or emergency primary inguinal hernia repair through any operative approach.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Compliance to audit standards described | A continuous 28-day period
  Mini-teams of up to five collaborators per data collection period will prospectively collect data on audit standards and confounding factors such as age, sex, BMI, ASA grade
Compliance to audit standards described | A continuous 28-day period
  Mini-teams of up to five collaborators per data collection period will prospectively collect data on audit standards and confounding factors such as BMI
Compliance to audit standards described | A continuous 28-day period
  Mini-teams of up to five collaborators per data collection period will prospectively collect data on audit standards and confounding factors such as ASA grade

SECONDARY OUTCOMES:
Number of patients with a 30-day follow-up | 30 days post surgery
  Considering there is no standard practice regarding if patients are evaluated at 30 days after surgery, whether in person or by phone, we establish to characterise this variation globally. Analysing the number of patients who had a phone follow-up and number of patients who did not have any follow up
30-day surgical site infection rates | 30 days post surgery
  Surgical site infection is defined at 30 days post-surgery using the Centers for Disease Control (CDC) definition of deep incisional or superficial incisional SSI
30-day reoperation rates | 30 days post surgery
  Re-operation within 30-days of the index operation
Number of patients re-admitted at 30-days | 30 days post surgery
  This will be related to postoperative complications that might require admission of patients and will be measured as number of patients readmitted at 30 days after surgery.
Number of patients who had a complication at 30 days, measured by Clavien-Dindo classification. | 30 days post surgery
  Adverse post-operative events within the follow-up period (30 days)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, Birmingham, United Kingdom